CLINICAL TRIAL: NCT05413174
Title: Contribution of Hypnosis in Guided Hepatic Biopsy
Brief Title: Contribution of Hypnosis in Guided Hepatic Biopsy (Ap-Hy-PBH)
Acronym: Ap-Hy-PBH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: APHP220124; 2022-A00008-35 (Other: ID-RCB Number)
Record Dates: First submitted 2022-05-20; First posted 2022-06-09 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Ultrasound-guided Hepatic Biopsy
Keywords: ultrasound-guided hepatic biopsy; radiology; hypnosis; anxiety; pain
MeSH Terms: conditions — Anxiety Disorders; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The Clinical Study Technician will then perform the 1:1 randomization. The randomization is automatically transmitted by email to the email of the radiology technician in charge of hypnosis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypnosis arm (Experimental): The experimental group will receive an hypnosis session during the ultrasound-guided hepatic biopsy.
  Interventions: Behavioral: Hypnoanalgésia
- Habitual Care (No Intervention): The control group will receive the usual medical management during the ultrasound-guided hepatic biopsy.

INTERVENTIONS:
Behavioral: Hypnoanalgésia — Use of Ericksonienne hypnosis in the medical field, aiming to dissociate the patient from the intervention in order to modify his or her perception of pain and limit anxiety.
  Ericksonienne hypnosis will use during ultrasound-guided biopsy in radiology ward.
  Arms: Hypnosis arm

SUMMARY:
The purpose of this study is to evaluate the contribution of hypnosis on the level of pain felt by the patient during ultrasound-guided hepatic biopsy, by comparing an intervention group (hypnosis) to a control group (routine and benevolent care).

Single-center randomized controlled trial.

DETAILED DESCRIPTION:
Hepatic Biopsy Puncture (HBP) is a very useful procedure for the assessment of chronic liver disease as well as in certain acute situations, and is also essential in oncology for the histological diagnosis of primary and secondary focal lesions. A study on the prevalence and characteristics of induced pain shows that it is a pain-generating procedure for 84% of patients and that the combination of anxiolytics and local anesthesia is insufficient. The effect of relaxing therapies was evaluated during percutaneous interventional radiology procedures. Anxiety and pain measured with visual analogue scales were significantly reduced in the group receiving support from sophrology and hypnosis . The mean evaluation of anxiety per procedure was 2.07 (95% CI, 1.48-2.82) in the group receiving relaxation therapy compared with 5.94 (95% CI, 4.62-7.22) in the other group. The mean level of pain felt was 1.83 (95% CI, 1.23-2.78) for the accompanied procedures versus 4.16 (95% CI, 2.53-6.04) without accompaniment. However, this study did not specifically look at percutaneous liver biopsy, and moreover the relaxation technique used was based on sophrology and not on an Ericksonian hypnosis approach.

Data concerning the use of hypnosis during percutaneous liver biopsies are limited to clinical cases, which report an absence of pain felt, including an observation in a patient who did not receive local anesthesia because of a history of allergy to Lidocaine.

Training in attentive and benevolent patient care already allows this type of procedure to be performed under good conditions in our department. This training of about one hour, carried out internally, does not require specific means. It would therefore seem useful to see what the impact is of using Ericksonian hypnosis, a recognized and risk-free technique which would require longer specific training for the staff and would represent a cost.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an indication for ultrasound-guided hepatic biopsy
* Over 18 years of age
* Affiliated to a social security system

Exclusion Criteria

* History of psychiatric pathology, psychotropic or anxiolytic treatments
* Refusal to participate.
* People who do not understand and/or speak French.
* People who are deaf
* Patients with impaired cognitive abilities, evaluated by the prescribing service
* Disorders of hemostasis against percutaneous approach
* Allergy to Lidocaine
* Patient under National Health Aids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2022-09-29 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-02 (Actual)

PRIMARY OUTCOMES:
Difference between groups of pain level during ultrasound-guided hepatic biopsy. | day 1
  maximal pain level feel (in a scale from 0 to 10, 0 means : no pain ; 10 means :maximal pain) during the process of ultrasound-guided hepatic biopsy.

SECONDARY OUTCOMES:
Difference between groups of anxiety level before the ultrasound-guided hepatic biopsy | day 1
  Maximal anxiety level feel (in a scale from 0 to 10, 0 means : no anxiety ; 10 means : maximal anxiety) before the process of ultrasound-guided hepatic biopsy.
Difference between groups of anxiety level during the ultrasound-guided hepatic biopsy | day 1
  Maximal anxiety level feel (in a scale from 0 to 10, 0 means : no anxiety ; 10 means : maximal anxiety) during the process of ultrasound-guided hepatic biopsy.
Difference between groups of pain level one hour after the ultrasound-guided hepatic biopsy. | day 1
  maximal pain level feel (in a scale from 0 to 10, 0 means : no pain ; 10 means :maximal pain) one hour following the ultrasound-guided hepatic biopsy.
Pain killer consumption | day 2
  Consumption of analgesic in the 24 hours following the ultrasound-guided hepatic biopsy (type of drug and cumulative doses).
Acceptability of another guided hepatic biopsy | day 2
  Acceptability of another ultrasound-guided hepatic biopsy (in a scale from 0 to 10, 0 means : totally refuse ; 10 means : accept without hesitation). This outcome will be collected 24 hours following the ultrasound-guided hepatic biopsy.

CONTACTS AND LOCATIONS:
Overall Officials: Véronique NITSCHE, RN, Study Director — APHP
Locations (1):
- AP-HP, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Eisenberg E, Konopniki M, Veitsman E, Kramskay R, Gaitini D, Baruch Y. Prevalence and characteristics of pain induced by percutaneous liver biopsy. Anesth Analg. 2003 May;96(5):1392-1396. doi: 10.1213/01.ANE.0000060453.74744.17. PMID 12707140
- [Background] Bertrand AS, Iannessi A, Buteau S, Jiang XY, Beaumont H, Grondin B, Baudin G. Effects of relaxing therapies on patient's pain during percutaneous interventional radiology procedures. Ann Palliat Med. 2018 Oct;7(4):455-462. doi: 10.21037/apm.2018.07.02. Epub 2018 Jul 20. PMID 30180736
- [Background] Adams PC, Stenn PG. Liver biopsy under hypnosis. J Clin Gastroenterol. 1992 Sep;15(2):122-4. doi: 10.1097/00004836-199209000-00008. PMID 1401822
- [Background] Kendrick C, Sliwinski J, Yu Y, Johnson A, Fisher W, Kekecs Z, Elkins G. Hypnosis for Acute Procedural Pain: A Critical Review. Int J Clin Exp Hypn. 2016;64(1):75-115. doi: 10.1080/00207144.2015.1099405. PMID 26599994
- [Background] Hauser W, Hagl M, Schmierer A, Hansen E. The Efficacy, Safety and Applications of Medical Hypnosis. Dtsch Arztebl Int. 2016 Apr 29;113(17):289-96. doi: 10.3238/arztebl.2016.0289. PMID 27173407
- [Background] Lindor KD, Bru C, Jorgensen RA, Rakela J, Bordas JM, Gross JB, Rodes J, McGill DB, Reading CC, James EM, Charboneau JW, Ludwig J, Batts KP, Zinsmeister AR. The role of ultrasonography and automatic-needle biopsy in outpatient percutaneous liver biopsy. Hepatology. 1996 May;23(5):1079-83. doi: 10.1002/hep.510230522. PMID 8621137
- [Background] Cadranel JF, Rufat P, Degos F. [Practices of transcutaneous liver biopsies in France. Results of a retrospective nationwide study]. Gastroenterol Clin Biol. 2001 Jan;25(1):77-80. French. PMID 11275620
- [Background] Alexander JA, Smith BJ. Midazolam sedation for percutaneous liver biopsy. Dig Dis Sci. 1993 Dec;38(12):2209-11. doi: 10.1007/BF01299897. PMID 8261822
- [Background] Castera L, Negre I, Samii K, Buffet C. Patient-administered nitrous oxide/oxygen inhalation provides safe and effective analgesia for percutaneous liver biopsy: a randomized placebo-controlled trial. Am J Gastroenterol. 2001 May;96(5):1553-7. doi: 10.1111/j.1572-0241.2001.03776.x. PMID 11374698
- [Background] Froehlich F, Lamy O, Fried M, Gonvers JJ. Practice and complications of liver biopsy. Results of a nationwide survey in Switzerland. Dig Dis Sci. 1993 Aug;38(8):1480-4. doi: 10.1007/BF01308607. PMID 8344104
- [Background] Faymonville ME, Laureys S, Degueldre C, DelFiore G, Luxen A, Franck G, Lamy M, Maquet P. Neural mechanisms of antinociceptive effects of hypnosis. Anesthesiology. 2000 May;92(5):1257-67. doi: 10.1097/00000542-200005000-00013. PMID 10781270
- [Result] Barat M, Ollivier C, Taibi L, Nitsche V, Sogni P, Soyer P, Parlati L, Dohan A, Abdoul H, Revel MP. Standard of care versus standard of care plus Ericksonian hypnosis for percutaneous liver biopsy: Results of a randomized control trial. Diagn Interv Imaging. 2025 Mar;106(3):93-97. doi: 10.1016/j.diii.2024.09.009. Epub 2024 Oct 2. PMID 39358154